CLINICAL TRIAL: NCT06424925
Title: Use of Artificial Intelligence (AI) for the Prediction of Clinical Outcomes Such as Death and Complications in Patients Hospitalized for COVID Pneumonia During the 4 Pandemic Waves at the ASST of Lecco.
Brief Title: Use of Artificial Intelligence (AI) to Predict Clinical Outcomes in Patients Hospitalized for COVID19 Pneumonia During the 4 Pandemic Waves
Acronym: AI COVID-19
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Ospedaliera di Lecco (Other)
Responsible Party: Principal Investigator, Stefania Piconi, Director of Infectious Diseases Unit, Azienda Ospedaliera di Lecco
Other Study IDs: AI COVID-19
Record Dates: First submitted 2024-05-21; First posted 2024-05-22 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — Artificial Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- COVID-19 1° wave: Hospitalized patients for COVID19 pneumonia during first wave (FEB-MAY 2020)
  Interventions: Other: Artificial intelligence for the prediction of clinical outcomes
- COVID-19 2° wave: Hospitalized patients for COVID19 pneumonia during the second wave (OCT-DEC 2020)
  Interventions: Other: Artificial intelligence for the prediction of clinical outcomes
- COVID-19 3° wave: Hospitalized patients for COVID19 pneumonia during the third wave (GEN-MAY 2021)
  Interventions: Other: Artificial intelligence for the prediction of clinical outcomes
- COVID-19 4° wave: Hospitalized patients for COVID19 pneumonia during the fourth wave (NOV 2021-MAR 2022)
  Interventions: Other: Artificial intelligence for the prediction of clinical outcomes

INTERVENTIONS:
Other: Artificial intelligence for the prediction of clinical outcomes — Use of artificial intelligence (AI) for the prediction of clinical outcomes such as death and complications in patients hospitalized for COVID pneumonia during the 4 pandemic waves

SUMMARY:
Predictive models can be applied in different areas, during the emergency of the COVID-19 pandemic, in fact, they have proven important in supporting health systems in planning strategic decisions and in formulating health policies for the containment of the disease.

The Covid-19 pandemic, in particular, has represented a real challenge for our healthcare system. In Italy, it was divided into four main waves, each characterized by different types of patients and different therapeutic approaches progressively improved based on new scientific evidence.

The objective is to carry out a study on the data of patients hospitalized for COVID-19 at the ASST of Lecco during all four pandemic waves, with different degrees of severity of illness, collecting the data of interest and applying it to they use artificial intelligence to identify recurring patterns of clinical outcome in terms of survival and secondary infectious complications, so as to build new reliable predictive statistical models that can be used to predict the outcome of the patients themselves.

The strong ambition of this project is that the application of artificial intelligence to data of such significant quantity can allow us to build valid statistical models which can then be hypothetically applied to any patient to predict, based on anamnestic characteristics, blood chemical parameters. at baseline and at the set treatment, the probability of survival and complications

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Hospitalization for COVID-19 pneumonia at ASST Lecco.

Exclusion Criteria:

* Hospitalization or finding of asymptomatic SARS CoV-2 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For each patient, information will be collected regarding:
  * Personal data (i.e. age, sex, nationality);
  * Date of hospitalization and discharge (or death)
  * Comorbidities;
  * Treatments undertaken for Covid19;
  * Possible vaccination for Covid19, date and number of doses;
  * Possible onset of secondary infections and/or complications;
  * Blood chemistry tests upon admission
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Construction of predictive models | 6 months
  Construction of predictive models to evaluate clinical outcomes such as death and/or onset of secondary infection based on the data collected relating to the 4 COVID-19 waves.

CONTACTS AND LOCATIONS:
Locations (1):
- Stefania Piconi, Lecco, Italy